CLINICAL TRIAL: NCT01250756
Title: A Phase 4, Randomized, Open-label Trial Evaluating the Safety, Tolerability, and Immunogenicity of DTaP Vaccine in Healthy Infants Given With a 7-valent Pneumococcal Conjugate Vaccine in Japan.
Brief Title: A Trial Evaluating a 7-valent Pneumococcal Conjugate Vaccine Given With Diphtheria, Tetanus, and Acellular Pertussis Vaccine (DTaP) in Healthy Japanese Infants.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B1841007; B1841007, 6107A1-4000
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Subjects
Keywords: vaccine; pneumococcal conjugate
MeSH Terms: interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Experimental
  Interventions: Biological: 7-pneumococcal conjugate vaccine (7vPnC); Biological: diphtheria, tetanus, and acellular pertussis vaccine (DTaP)
- 2 (Experimental): Active comparator
  Interventions: Biological: DTaP

INTERVENTIONS:
Biological: 7-pneumococcal conjugate vaccine (7vPnC) — 0.5 mL per dose, 4 doses
  Arms: 1
Biological: diphtheria, tetanus, and acellular pertussis vaccine (DTaP) — 0.5 mL per dose, 4 doses
  Arms: 1
Biological: DTaP — 0.5 mL per dose, 4 doses
  Arms: 2

SUMMARY:
Subjects will be randomly assigned to 1 of 2 groups to receive the following vaccines: Group 1: 7-valent pneumococcal conjugate vaccine (7vPnC) and diphtheria, tetanus, and accelular pertussis vaccine (DTaP), Group 2: DTaP alone. Group 2 subjects will also receive catch-up doses of 7vPnC. The study vaccines will be open-label. The main purpose of the study is to demonstrate that the immune responses as measured by serum antibody responses to diphtheria toxin, tetanus toxin, pertussis toxin (PT) and filamentous haemagglutinin (FHA) induced by DTaP given concomitantly with 7vPnC are comparable to the immune responses induced by DTaP given alone. In addition, the study aims to evaluate the side effects (safety profile) after vaccination of 7vPnC when given with DTaP in healthy Japanese infants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 to 6 months (defined as the first day the subject is 3 months of age to the last day the subject is 6 months of age) at time of enrollment.
* Available for entire study period and whose parent/legal guardian can be reached by telephone.
* Healthy infant as determined by medical history, physical examination, and judgment of the investigator.

Exclusion Criteria:

* Previous vaccination with licensed or investigational pneumococcal, diphtheria, tetanus, or pertussis vaccines.
* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate any type of injection.
* History of culture-proven invasive disease caused by S pneumoniae (eg, meningitis, bacteremia, osteomyelitis, arthritis).
* Subjects who are direct descendants (child, grandchild) of investigational site staff members or subjects who are direct descendants (child, grandchild) of Pfizer employees directly involved in the conduct of the trial.

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 321 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Japan (18):
  - Tsubaki Children's Clinic, Chiba, Chiba
  - Sotobo Children's Clinic, Isumi, Chiba
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Kiyomatsu Childrens Clinic, Fukuoka, Fukuoka
  - National Hospital Organization Fukuoka National Hospital, Fukuoka, Fukuoka
  - Shindo Children's Clinic, Fukuoka, Fukuoka
  - Takasaki Clinic Pedatrics and Child Health, Fukuoka, Fukuoka
  - Yamashita Pediatrics Clinic, Itoshima, Fukuoka
  - Yokoyama Children's Clinic, Kasuga, Fukuoka
  - Furuta Children's Clinic, Sapporo, Hokkaido
  - Tenshi Hospital, Sapporo, Hokkaido
  - Watanabe Pediatric Allergy Clinic, Sapporo, Hokkaido
  - Yamanaka Tatsuru Pediatrics, Sapporo, Hokkaido
  - Matsuda Pediatrics Clinic, Kuwana, Mie-ken
  - Kawasaki Medical School, Department of Pediatrics, Kurashiki, Okayama-ken
  - Momotaro Clinic, Okayama, Okayama-ken
  - Hug Hug Kids Clinic, Toyonaka, Osaka
  - Shibuya Clinic, Kumagaya, Saitama

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1841007&StudyName=A%20Trial%20Evaluating%20a%207-valent%20Pneumococcal%20Conjugate%20Vaccine%20Given%20with%20Diphtheria%2C%20Tetanus%2C%20and%20Acellular%20Pertussis%20Vaccine%20%28DTaP%29%20

RESULTS

PARTICIPANT FLOW:
Groups:
- 7vPnC + DTaP: Participants at 3 to 6 months of age received a single 0.5 milliliter (mL) dose of 7-valent pneumococcal conjugate vaccine (7vPnC) subcutaneously followed by 2 single 0.5 mL doses of 7vPnC subcutaneously, 4 to 8 weeks after each previous dose (infant series) and a single 0.5 mL dose of 7vPnC subcutaneously at 12 to 15 months of age (toddler dose). A single 0.5 mL dose of diphtheria, tetanus, and acellular pertussis vaccine (DTaP) subcutaneously administered concomitantly with each 7vPnC dose.
- DTaP (Catch-up 7vPnC): Participants at 3 to 6 months of age received a single 0.5 mL DTaP dose subcutaneously followed by 2 single 0.5 mL DTaP doses subcutaneously, 4 to 8 weeks after each previous dose (infant series). Four to 6 weeks post-infant series, 2 single catch-up (CU) doses of 7vPnC (Prevenar) were administered subcutaneously, 4 to 6 weeks apart. A single 0.5 mL DTaP dose subcutaneously at 12 to 15 months of age (toddler dose) followed by a single CU dose of 7vPnC (Prevenar) subcutaneously 4 to 6 weeks post-toddler dose.
Period: Infant Series
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Started | 161 | 160
Vaccinated Dose 1 | 159 | 158
Vaccinated Dose 2 | 147 | 157
Vaccinated Dose 3 | 133 | 155
Completed | 133 | 153
Not Completed | 28 | 7
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Randomized, Not Vaccinated | 2 | 2
Not completed — Other | 22 | 0
Period: After Infant Series
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Started | 133 | 153
Completed | 122 | 149
Not Completed | 11 | 4
Not completed — Adverse Event | 5 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Other | 2 | 1
Period: Toddler Dose
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Started | 122 | 149
Completed | 122 | 148
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: After Toddler Dose
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Started | 0 | 148
Completed | 0 | 147
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC) | Total
Number analyzed (Participants) | 161 | 160 | 321
Age Continuous [Mean (Standard Deviation); unit: months] | 3.8 (0.91) | 3.9 (0.94) | 3.9 (0.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 82 | 162
  Male | 81 | 78 | 159

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Diphtheria Toxoid, Tetanus Toxoid, and Pertussis Antigens 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody level along with the corresponding 95% confidence interval (CI) were presented. Exact 2-sided CI based on the observed proportion of participants. Predefined antibody levels were 0.1 International Units/mL (IU/mL) for diphtheria, 0.01 IU/mL for tetanus, 5 Enzyme-linked Immunosorbent Assay (ELISA) units/mL (EU/mL) for pertussis toxoid (PT), and 5 EU/mL for filamentous hemagglutinin (FHA).
Time Frame: 1 month after the infant series
Population: Evaluable infant immunogenicity population: eligible participants who received the vaccine to which they were randomized at all 3 doses, had blood drawn within the protocol-specified time frames, had at least 1 valid, determinate assay result for proposed analysis, received no prohibited vaccines, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 132 | 149
Percentage of participants
  Diphtheria | 100.0 [97.2 to 100.0] | 100.0 [97.6 to 100.0]
  Tetanus | 100.0 [97.2 to 100.0] | 100.0 [97.6 to 100.0]
  Pertussis toxoid (PT) | 100.0 [97.2 to 100.0] | 100.0 [97.6 to 100.0]
  Filamentous hemagglutinin (FHA) | 100.0 [97.2 to 100.0] | 100.0 [97.6 to 100.0]

2. Primary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Diphtheria and Tetanus Antibody 1 Month After the Infant Series
Description: Geometric mean concentrations (GMCs) were measured in IU/mL and corresponding 2-sided 95% confidence interval (CI) were evaluated for diphtheria and tetanus antibodies.
Time Frame: 1 month after the infant series
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 132 | 149
IU/mL
  Diphtheria | 1.38 [1.27 to 1.49] | 0.99 [0.91 to 1.09]
  Tetanus | 1.91 [1.69 to 2.16] | 2.05 [1.83 to 2.29]

3. Primary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Acellular Pertussis Antibody 1 Month After the Infant Series
Description: GMCs were measured in EU/mL and corresponding 2-sided 95% CI were evaluated for PT and FHA antibodies.
Time Frame: 1 month after the infant series
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 132 | 149
EU/mL
  Pertussis toxoid (PT) | 76.79 [70.81 to 83.28] | 83.56 [77.54 to 90.05]
  Filamentous hemagglutinin (FHA) | 72.89 [65.80 to 80.74] | 77.85 [71.01 to 85.35]

4. Primary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Level Greater Than or Equal to (>=) 0.35 Microgram Per Milliliter (Mcg/mL) 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold >=0.35 mcg/mL along with the corresponding 95% CI for the 7 pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F and 23F) were presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: 1 month after the infant series
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 7vPnC + DTaP
Number analyzed (Participants) | 132
Percentage of participants
  4 | 100.0 [97.2 to 100.0]
  6B | 99.2 [95.9 to 100.0]
  9V | 100.0 [97.2 to 100.0]
  14 | 99.2 [95.9 to 100.0]
  18C | 99.2 [95.8 to 100.0]
  19F | 97.7 [93.5 to 99.5]
  23F | 98.5 [94.6 to 99.8]

5. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Infant Series
Description: Antibody geometric mean concentrations (GMCs) for 7 pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) were presented. GMC and corresponding 2-sided 95% CI were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after the infant series
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 7vPnC + DTaP
Number analyzed (Participants) | 132
mcg/mL
  4 | 11.82 [10.50 to 13.31]
  6B | 4.23 [3.61 to 4.97]
  9V | 5.96 [5.37 to 6.62]
  14 | 16.61 [14.66 to 18.81]
  18C | 5.48 [4.76 to 6.31]
  19F | 8.85 [7.54 to 10.40]
  23F | 4.17 [3.54 to 4.91]

6. Secondary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Diphtheria Toxoid, Tetanus Toxoid, and Pertussis Antigens 1 Month After the Toddler Dose
Description: Percentage of participants achieving predefined antibody level along with the corresponding 95% CI were presented. Exact 2-sided CI based on the observed proportion of participants. Predefined antibody levels were 0.1 IU/mL for diphtheria, 0.01 IU/mL for tetanus, 5 EU/mL for PT, and 5 EU/mL for FHA.
Time Frame: 1 month after the toddler dose
Population: Evaluable toddler immunogenicity set: eligible participants who received vaccine to which they were randomized at all 4 doses, had blood drawn within protocol-specified time, had at least 1 valid, determinate assay result after toddler dose for analysis, received no prohibited vaccines, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 121 | 146
Percentage of participants
  Diphtheria | 100.0 [97.0 to 100.0] | 100.0 [97.5 to 100.0]
  Tetanus | 100.0 [97.0 to 100.0] | 100.0 [97.5 to 100.0]
  Pertussis toxoid (PT) | 100.0 [97.0 to 100.0] | 100.0 [97.5 to 100.0]
  Filamentous hemagglutinin (FHA) | 100.0 [97.0 to 100.0] | 100.0 [97.5 to 100.0]

7. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Diphtheria and Tetanus Antibody 1 Month After the Toddler Dose
Description: GMCs were measured in IU/mL and corresponding 2-sided 95% CI were evaluated for diphtheria and tetanus antibodies.
Time Frame: 1 month after the toddler dose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 121 | 146
IU/mL
  Diphtheria | 2.56 [2.35 to 2.78] | 2.14 [1.94 to 2.35]
  Tetanus | 2.53 [2.26 to 2.82] | 3.04 [2.74 to 3.38]

8. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Acellular Pertussis Antibody 1 Month After the Toddler Dose
Description: GMCs were measured in EU/mL and corresponding 2-sided 95% CI were evaluated for PT and FHA antibodies.
Time Frame: 1 month after the toddler dose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 121 | 146
EU/mL
  PT | 106.54 [96.10 to 118.12] | 130.62 [119.60 to 142.65]
  FHA | 120.99 [109.75 to 133.39] | 145.38 [132.41 to 159.63]

9. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Level >=0.35 Mcg/mL 1 Month After the Toddler Dose
Description: as for outcome 4
Time Frame: 1 month after the toddler dose
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 7vPnC + DTaP
Number analyzed (Participants) | 121
Percentage of participants
  4 | 100.0 [97.0 to 100.0]
  6B | 100.0 [97.0 to 100.0]
  9V | 100.0 [97.0 to 100.0]
  14 | 100.0 [97.0 to 100.0]
  18C | 99.2 [95.5 to 100.0]
  19F | 99.2 [95.5 to 100.0]
  23F | 100.0 [97.0 to 100.0]

10. Secondary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Toddler Dose
Description: Antibody GMCs for 7 pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) were presented. GMC and corresponding 2-sided 95% CIs were evaluated. GMs were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after the toddler dose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 7vPnC + DTaP
Number analyzed (Participants) | 121
mcg/mL
  4 | 12.15 [10.35 to 14.26]
  6B | 10.66 [8.96 to 12.68]
  9V | 6.43 [5.57 to 7.42]
  14 | 15.83 [13.81 to 18.14]
  18C | 6.53 [5.49 to 7.76]
  19F | 9.70 [8.15 to 11.56]
  23F | 10.17 [8.58 to 12.07]

11. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Pneumococcal Antibodies From Pretoddler Dose to 1 Month After the Toddler Dose
Description: Geometric mean fold rises (GMFRs) for the 7 pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) from prevaccination to 1 month postvaccination were computed using the logarithmically transformed assay results. CI for the GMFRs were back transformations of a CI based on the Student t distribution for the logarithmically transformed assay results.
Time Frame: Pre-toddler dose, 1 month after the toddler dose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | 7vPnC + DTaP
Number analyzed (Participants) | 121
Fold Rise
  4 | 6.74 [5.75 to 7.90]
  6B | 5.89 [5.09 to 6.81]
  9V | 4.34 [3.81 to 4.93]
  14 | 3.63 [3.22 to 4.09]
  18C | 6.90 [6.06 to 7.85]
  19F | 6.37 [5.35 to 7.59]
  23F | 8.10 [7.01 to 9.35]

12. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Level >=0.35 Mcg/mL 1 Month After Catch-up Dose 3
Description: as for outcome 4
Time Frame: 1 month after the catch-up dose 3
Population: Catch-up immunogenicity population: eligible participants who received the vaccine to which they were randomized at all 3 catch-up doses, had blood drawn within the protocol-specified time frames, had at least 1 valid, determinate assay result for proposed analysis, received no prohibited vaccines, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 148
Percentage of participants
  4 | 100.0 [97.5 to 100.0]
  6B | 99.3 [96.3 to 100.0]
  9V | 100.0 [97.5 to 100.0]
  14 | 100.0 [97.5 to 100.0]
  18C | 99.3 [96.3 to 100.0]
  19F | 100.0 [97.5 to 100.0]
  23F | 99.3 [96.3 to 100.0]

13. Secondary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After Catch-up Dose 3
Description: Antibody GMCs for 7 pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) were presented. GMC and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after the catch-up dose 3
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 148
mcg/mL
  4 | 6.63 [5.91 to 7.44]
  6B | 4.30 [3.75 to 4.93]
  9V | 3.48 [3.12 to 3.89]
  14 | 11.55 [10.30 to 12.95]
  18C | 3.10 [2.69 to 3.57]
  19F | 5.16 [4.45 to 5.99]
  23F | 4.41 [3.78 to 5.14]

14. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Infant Series Dose 1 (3 to 6 Months of Age)
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Erythema and induration were scaled as Any (erythema and induration present); Mild (0.5 to 2.0 centimeters [cm]); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category. Injection site being evaluated for local reactions was 7vPnC injection site in the 7vPnC+DTaP group, and DTaP injection site in the DTaP (Catch-up 7vPnC) group.
Time Frame: Within 7 days after Dose 1 of the infant series
Population: Safety population included all participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any local reaction. 'n'=participants reporting yes for at least 1 day or no for all days for the specified local reaction for each group, respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 152 | 154
Percentage of participants
  Erythema-Any (n= 152, 152) | 57.2 | 14.5
  Erythema-Mild (n= 152, 151) | 52.6 | 12.6
  Erythema-Moderate (n= 148, 152) | 14.9 | 2.0
  Erythema-Severe (n= 148, 151) | 0.0 | 0.0
  Induration-Any (n= 149, 153) | 40.3 | 7.8
  Induration-Mild (n= 149, 153) | 38.3 | 7.8
  Induration-Moderate (n= 148, 151) | 10.1 | 0.0
  Induration-Severe (n= 148, 151) | 0.0 | 0.0
  Tenderness-Any (n= 148, 151) | 12.2 | 0.7
  Tenderness-Significant (n= 148, 151) | 0.0 | 0.0
  Any local reaction (n= 152, 154) | 66.4 | 15.6

15. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Infant Series Dose 2 (4 to 8 Months of Age)
Description: as for outcome 14
Time Frame: Within 7 days after Dose 2 of the infant series
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 143 | 151
Percentage of participants
  Erythema-Any (n= 142, 150) | 64.1 | 39.3
  Erythema-Mild (n= 142, 150) | 58.5 | 33.3
  Erythema-Moderate (n= 134, 147) | 32.1 | 6.8
  Erythema-Severe (n= 133, 147) | 0.0 | 0.0
  Induration-Any (n= 137, 150) | 51.8 | 30.0
  Induration-Mild (n= 137, 150) | 49.6 | 28.7
  Induration-Moderate (n= 134, 148) | 23.9 | 6.8
  Induration-Severe (n= 133, 147) | 0.0 | 0.0
  Tenderness-Any (n= 133, 147) | 7.5 | 4.1
  Tenderness-Significant (n= 133, 147) | 0.0 | 0.0
  Any local reaction (n= 143, 151) | 69.2 | 45.0

16. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Infant Series Dose 3 (5 to 10 Months of Age)
Description: as for outcome 14
Time Frame: Within 7 days after Dose 3 of the infant series
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 126 | 145
Percentage of participants
  Erythema-Any (n= 123, 144) | 52.8 | 30.6
  Erythema-Mild (n= 123, 143) | 46.3 | 28.0
  Erythema-Moderate (n= 120, 139) | 20.0 | 5.8
  Erythema-Severe (n= 118, 138) | 0.0 | 0.0
  Induration-Any (n= 124, 144) | 44.4 | 19.4
  Induration-Mild (n= 124, 144) | 42.7 | 19.4
  Induration-Moderate (n= 119, 139) | 11.8 | 2.2
  Induration-Severe (n= 118, 138) | 0.0 | 0.0
  Tenderness-Any (n= 119, 138) | 5.0 | 3.6
  Tenderness-Significant (n= 118, 138) | 0.0 | 0.0
  Any local reaction (n= 126, 145) | 61.1 | 33.1

17. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Toddler Dose (12 to 15 Months of Age)
Description: as for outcome 14
Time Frame: Within 7 days after the toddler dose
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 110 | 138
Percentage of participants
  Erythema-Any (n= 108, 137) | 51.9 | 32.1
  Erythema-Mild (n= 106, 137) | 48.1 | 28.5
  Erythema-Moderate (n= 102, 134) | 23.5 | 7.5
  Erythema-Severe (n= 98, 133) | 0.0 | 0.0
  Induration-Any (n= 108, 137) | 42.6 | 23.4
  Induration-Mild (n= 108, 137) | 40.7 | 19.7
  Induration-Moderate (n= 99, 133) | 16.2 | 6.8
  Induration-Severe (n= 98, 133) | 0.0 | 0.0
  Tenderness-Any (n= 99, 136) | 11.1 | 4.4
  Tenderness-Significant (n= 98, 133) | 0.0 | 0.0
  Any local reaction (n= 110, 138) | 56.4 | 39.1

18. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Post Infant Series Catch-up Dose 1 (6 to 11.5 Months of Age)
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Erythema and induration were scaled as Any (erythema and induration present); Mild (0.5 to 2.0 centimeters [cm]); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category. Injection site being evaluated for local reactions was catch-up 7vPnC injection site in the DTaP (Catch-up 7vPnC) group.
Time Frame: Within 7 days after Catch-up Dose 1
Population: Safety population included all participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any local reaction. 'n'=participants reporting yes for at least 1 day or no for all days for the specified local reaction.
Measure: Number; unit: Percentage of participants
Arm/Group | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 141
Percentage of participants
  Erythema-Any (n= 139) | 51.8
  Erythema-Mild (n= 139) | 45.3
  Erythema-Moderate (n= 136) | 10.3
  Erythema-Severe (n= 135) | 0.0
  Induration-Any (n= 138) | 34.8
  Induration-Mild (n= 138) | 32.6
  Induration-Moderate (n= 135) | 8.1
  Induration-Severe (n= 135) | 0.0
  Tenderness-Any (n= 136) | 8.1
  Tenderness-Significant (n= 135) | 0.0
  Any local reaction (n= 141) | 54.6

19. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Post Infant Series Catch-up Dose 2 (7 to 13 Months of Age)
Description: as for outcome 18
Time Frame: Within 7 days after Catch-up Dose 2
Population: as for outcome 18
Measure: Number; unit: Percentage of participants
Arm/Group | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 145
Percentage of participants
  Erythema-Any (n= 144) | 50.7
  Erythema-Mild (n= 144) | 45.1
  Erythema-Moderate (n= 140) | 13.6
  Erythema-Severe (n= 138) | 0.0
  Induration-Any (n= 144) | 32.6
  Induration-Mild (n= 143) | 30.1
  Induration-Moderate (n= 140) | 15.0
  Induration-Severe (n= 138) | 0.0
  Tenderness-Any (n= 139) | 5.0
  Tenderness-Significant (n= 138) | 0.0
  Any local reaction (n= 145) | 55.2

20. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Post Infant Series Catch-up Dose 3 (13 to16.5 Months of Age)
Description: as for outcome 18
Time Frame: Within 7 days after Catch-up Dose 3
Population: as for outcome 18
Measure: Number; unit: Percentage of participants
Arm/Group | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 137
Percentage of participants
  Erythema-Any (n= 134) | 32.1
  Erythema-Mild (n= 133) | 27.1
  Erythema-Moderate (n= 131) | 9.9
  Erythema-Severe (n= 130) | 0.0
  Induration-Any (n= 134) | 27.6
  Induration-Mild (n= 133) | 24.8
  Induration-Moderate (n= 131) | 9.9
  Induration-Severe (n= 130) | 0.0
  Tenderness-Any (n= 132) | 6.8
  Tenderness-Significant (n= 130) | 0.0
  Any local reaction (n= 137) | 40.9

21. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Infant Series Dose 1 (3 to 6 Months of Age)
Description: Systemic events (any fever >= 37.5 degrees Celsius [C], decreased appetite, irritability, increased sleep, decreased sleep, and hives [urticaria]), were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after Dose 1 of the infant series
Population: Safety population included all participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any systemic event. 'n'=participants reporting yes for at least 1 day or no for all days for specified systemic reaction for each group, respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 154 | 153
Percentage of participants
  Fever >=37.5 but =<39 degrees C(n=149,152) | 18.8 | 15.8
  Fever >39 but =<40.0 degrees C(n=148,151) | 2.0 | 2.0
  Fever >40 degrees C(n=148,151) | 0.0 | 0.0
  Decreased appetite(n=148,151) | 8.8 | 7.9
  Irritability(n=151,151) | 15.2 | 9.3
  Increased sleep(n=150,153) | 32.0 | 25.5
  Decreased sleep(n=151,151) | 16.6 | 15.2
  Hives (urticaria)(n=148,151) | 1.4 | 0.7
  Antipyretic medication to treat symptom(n=148,151) | 1.4 | 1.3
  Any systemic event(n=154,153) | 57.8 | 48.4

22. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Infant Series Dose 2 (4 to 8 Months of Age)
Description: as for outcome 21
Time Frame: Within 7 days after Dose 2 of the infant series
Population: as for outcome 21
Measure: Number; unit: Percentage of participants
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 142 | 153
Percentage of participants
  Fever >=37.5 but =<39 degrees C(n=138,149) | 25.4 | 15.4
  Fever >39 but =<40.0 degrees C(n=135,147) | 2.2 | 0.0
  Fever >40 degrees C(n=133,147) | 0.0 | 0.7
  Decreased appetite(n=135,147) | 11.9 | 5.4
  Irritability(n=134,149) | 19.4 | 12.1
  Increased sleep(n=136,148) | 19.1 | 12.8
  Decreased sleep(n=140,151) | 17.1 | 15.2
  Hives (urticaria)(n=133,147) | 3.0 | 0.0
  Antipyretic medication to treat symptom(n=134,147) | 2.2 | 2.0
  Any systemic event(n=142,153) | 53.5 | 38.6

23. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Infant Series Dose 3 (5 to 10 Months of Age)
Description: as for outcome 21
Time Frame: Within 7 days after Dose 3 of the infant series
Population: as for outcome 21
Measure: Number; unit: Percentage of participants
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 122 | 143
Percentage of participants
  Fever >=37.5 but =<39 degrees C(n=120,141) | 19.2 | 14.9
  Fever >39 but =<40.0 degrees C(n=118,138) | 1.7 | 0.7
  Fever >40 degrees C(n=118,138) | 0.0 | 0.0
  Decreased appetite(n=119,138) | 8.4 | 6.5
  Irritability(n=118,139) | 10.2 | 7.2
  Increased sleep(n=119,141) | 16.0 | 18.4
  Decreased sleep(n=120,140) | 6.7 | 14.3
  Hives (urticaria)(n=119,138) | 1.7 | 0.0
  Antipyretic medication to treat symptom(n=119,138) | 1.7 | 2.2
  Any systemic event(n=122,143) | 39.3 | 36.4

24. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Toddler Dose (12 to 15 Months of Age)
Description: as for outcome 21
Time Frame: Within 7 days after the toddler dose
Population: as for outcome 21
Measure: Number; unit: Percentage of participants
Arm/Group | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 108 | 138
Percentage of participants
  Fever >=37.5 but =<39 degrees C(n=103,135) | 34.0 | 22.2
  Fever >39 but =<40.0 degrees C(n=99,132) | 5.1 | 2.3
  Fever >40 degrees C(n=98,132) | 1.0 | 0.0
  Decreased appetite(n=100,133) | 9.0 | 8.3
  Irritability(n=100,134) | 17.0 | 9.7
  Increased sleep(n=103,135) | 20.4 | 15.6
  Decreased sleep(n=101,133) | 10.9 | 7.5
  Hives (urticaria)(n=98,133) | 1.0 | 0.8
  Antipyretic medication to treat symptom(n=98,133) | 4.1 | 4.5
  Any systemic event(n=108,138) | 52.8 | 39.9

25. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Post Infant Series Catch-up Dose 1 (6 to 11.5 Months of Age)
Description: as for outcome 21
Time Frame: Within 7 days after Catch-up Dose 1
Population: Safety population included all participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any systemic event. 'n'=participants reporting yes for at least 1 day or no for all days for specified systemic reaction.
Measure: Number; unit: Percentage of participants
Arm/Group | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 139
Percentage of participants
  Fever >=37.5 but =<39 degrees C(n=139) | 32.4
  Fever >39 but =<40.0 degrees C(n=135) | 2.2
  Fever >40 degrees C(n=135) | 0.0
  Decreased appetite(n=136) | 8.1
  Irritability(n=136) | 12.5
  Increased sleep(n=136) | 17.6
  Decreased sleep(n=136) | 11.8
  Hives (urticaria)(n=135) | 0.7
  Antipyretic medication to treat symptom(n=136) | 5.9
  Any systemic event(n=139) | 49.6

26. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Post Infant Series Catch-up Dose 2 (7 to 13 Months of Age)
Description: as for outcome 21
Time Frame: Within 7 days after Catch-up Dose 2
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 141
Percentage of participants
  Fever >=37.5 but =<39 degrees C(n=140) | 32.1
  Fever >39 but =<40.0 degrees C(n=138) | 5.1
  Fever >40 degrees C(n=138) | 0.7
  Decreased appetite(n=138) | 10.9
  Irritability(n=138) | 11.6
  Increased sleep(n=138) | 15.9
  Decreased sleep(n=139) | 10.1
  Hives (urticaria)(n=138) | 2.2
  Antipyretic medication to treat symptom(n=138) | 5.1
  Any systemic event(n=141) | 47.5

27. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Post Infant Series Catch-up Dose 3 (13 to 16.5 Months of Age)
Description: as for outcome 21
Time Frame: Within 7 days after Catch-up Dose 3
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 136
Percentage of participants
  Fever >=37.5 but =<39 degrees C(n=134) | 26.9
  Fever >39 but =<40.0 degrees C(n=130) | 0.8
  Fever >40 degrees C(n=130) | 0.0
  Decreased appetite(n=130) | 6.2
  Irritability(n=131) | 9.2
  Increased sleep(n=131) | 10.7
  Decreased sleep(n=131) | 6.9
  Hives (urticaria)(n=131) | 0.8
  Antipyretic medication to treat symptom(n=130) | 1.5
  Any systemic event(n=136) | 39.0

ADVERSE EVENTS:
Time Frame: AEs/SAEs: recorded from signing of informed consent form to completion of study. Participants recorded prespecified AEs in electronic diary:local reactions; systemic events; use of antipyretic medication (up to 7 days after each vaccine dose).
Description: Safety population: participants who receive at least 1 dose of study vaccine. SAEs and AEs were grouped by system organ class and summarized. AEs included solicited AEs collected in electronic diary (local and systemic reactions; systematic assessment) and unsolicited events collected on case report form at each visit (nonsystematic assessment).
Groups:
- 7vPnC + DTaP - Infant Series: Participants who received 3 single 0.5 mL doses of 7vPnC subcutaneously 4 to 8 weeks apart along with 3 single 0.5 mL doses of DTaP subcutaneously (infant series), assessed from Infant Dose 1 through the blood draw 28 to 42 days post-infant series.
- DTaP (Catch-up 7vPnC)- Infant Series: Participants who received 3 single 0.5 mL DTaP doses subcutaneously 4 to 8 weeks apart (infant series) followed by 2 single catch-up (CU) doses, CU Dose 1 and CU Dose 2 (separated by 4 to 6 weeks), of 7vPnC (Prevenar) 4 to 6 weeks post-infant series, assessed from Infant Dose 1 through the CU Dose 1.
- 7vPnC + DTaP - After the Infant Series: Participants who received 3 single 0.5 mL doses of 7vPnC subcutaneously 4 to 8 weeks apart along with 3 single 0.5 mL doses of DTaP subcutaneously (infant series), assessed after the infant series blood draw to the toddler dose.
- DTaP (Catch-up 7vPnC) - After the Infant Series: Participants who received 3 single 0.5 mL DTaP doses subcutaneously 4 to 8 weeks apart (infant series) followed by 2 single catch-up (CU) doses, CU Dose 1 and CU Dose 2 (separated by 4 to 6 weeks), of 7vPnC (Prevenar) 4 to 6 weeks post-infant series, assessed after CU Dose 1 to the toddler dose.
- 7vPnC + DTaP - Toddler Dose: Participants who received a single 0.5 mL dose of 7vPnC subcutaneously (toddler dose) along with 0.5 mL dose of DTaP subcutaneously, assessed from the toddler dose through the blood draw 28 to 42 days post-toddler dose.
- DTaP (Catch-up 7vPnC) - Toddler Dose: Participants who received a single 0.5 mL DTaP dose subcutaneously (toddler dose) followed by a single catch-up (CU) dose (CU Dose 3) of 7vPnC (Prevenar) 4 to 6 weeks after toddler dose; assessed from toddler dose through the CU Dose 3.
- DTaP (Catch-up 7vPnC) - After the Toddler Dose: Participants who received a single 0.5 mL DTaP dose subcutaneously (toddler dose) followed by a single catch-up (CU) dose (CU Dose 3) of 7vPnC (Prevenar) 4 to 6 weeks after toddler dose; assessed after the CU Dose 3 to 28 to 42 days post-CU Dose 3.
Arm/Group | 7vPnC + DTaP - Infant Series | DTaP (Catch-up 7vPnC)- Infant Series | 7vPnC + DTaP - After the Infant Series | DTaP (Catch-up 7vPnC) - After the Infant Series | 7vPnC + DTaP - Toddler Dose | DTaP (Catch-up 7vPnC) - Toddler Dose | DTaP (Catch-up 7vPnC) - After the Toddler Dose
Serious Adverse Events (participants affected / at risk) | 3/159 | 7/158 | 10/159 | 7/158 | 0/122 | 4/149 | 1/149
Other Adverse Events (participants affected / at risk) | 123/159 | 126/158 | 20/159 | 129/158 | 72/122 | 96/149 | 85/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 7vPnC + DTaP - Infant Series (N=159) | DTaP (Catch-up 7vPnC)- Infant Series (N=158) | 7vPnC + DTaP - After the Infant Series (N=159) | DTaP (Catch-up 7vPnC) - After the Infant Series (N=158) | 7vPnC + DTaP - Toddler Dose (N=122) | DTaP (Catch-up 7vPnC) - Toddler Dose (N=149) | DTaP (Catch-up 7vPnC) - After the Toddler Dose (N=149)
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis adenovirus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 4 | 2 | 0 | 1 | 1
Infantile asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Kawasaki's disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 7vPnC + DTaP - Infant Series (N=159) | DTaP (Catch-up 7vPnC)- Infant Series (N=158) | 7vPnC + DTaP - After the Infant Series (N=159) | DTaP (Catch-up 7vPnC) - After the Infant Series (N=158) | 7vPnC + DTaP - Toddler Dose (N=122) | DTaP (Catch-up 7vPnC) - Toddler Dose (N=149) | DTaP (Catch-up 7vPnC) - After the Toddler Dose (N=149)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 6 | 14 | 0 | 9 | 1 | 4 | 2
Eye discharge (Eye disorders) | 3 | 3 | 0 | 2 | 1 | 0 | 2
Keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 8 | 8 | 0 | 6 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 9 | 1 | 8 | 6 | 6 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0
Vaccination site erythema (General disorders) | 5 | 10 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 0 | 0 | 4 | 0 | 1 | 0
Vaccination site induration (General disorders) | 1 | 4 | 0 | 2 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vaccination site swelling (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 2 | 1 | 6 | 6 | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 49 | 59 | 1 | 63 | 27 | 43 | 42
Upper respiratory tract infection (Infections and infestations) | 35 | 22 | 5 | 27 | 17 | 19 | 10
Gastroenteritis (Infections and infestations) | 19 | 12 | 0 | 13 | 2 | 4 | 8
Influenza (Infections and infestations) | 16 | 12 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 10 | 11 | 0 | 17 | 11 | 12 | 9
Exanthema subitum (Infections and infestations) | 6 | 13 | 0 | 21 | 2 | 7 | 4
Gastroenteritis viral (Infections and infestations) | 7 | 3 | 0 | 2 | 0 | 0 | 1
Varicella (Infections and infestations) | 5 | 3 | 0 | 2 | 2 | 3 | 2
Impetigo (Infections and infestations) | 2 | 5 | 0 | 2 | 0 | 1 | 1
Otitis media (Infections and infestations) | 5 | 2 | 0 | 9 | 4 | 2 | 2
Respiratory syncytial virus infection (Infections and infestations) | 2 | 5 | 0 | 0 | 2 | 0 | 0
Bronchiolitis (Infections and infestations) | 5 | 1 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 5 | 0 | 0 | 0 | 0 | 4
Otitis media acute (Infections and infestations) | 0 | 5 | 0 | 4 | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 3 | 0 | 1 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 3 | 1
Gastroenteritis rotavirus (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 1 | 0
Adenovirus infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Genital candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 0 | 11 | 4 | 6 | 2
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucocutaneous candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal scalded skin syndrome (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 3 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 26 | 22 | 2 | 4 | 2 | 3 | 5
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 16 | 13 | 1 | 13 | 7 | 2 | 4
Eczema infantile (Skin and subcutaneous tissue disorders) | 6 | 8 | 1 | 1 | 0 | 0 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 5 | 4 | 0 | 1 | 1 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 6 | 1 | 2 | 1 | 1 | 1
Heat rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 16 | 2 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 | 0 | 3 | 2 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3 | 0 | 2 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infantile asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis perennial (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergy to animal (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Herpangina (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida nappy rash (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis adenovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Any) (Skin and subcutaneous tissue disorders) | 87/152 | 22/152 | 0/0 | 72/139 | 56/108 | 44/137 | 0/0 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose
Erythema (Any) (Skin and subcutaneous tissue disorders) | 91/142 | 59/150 | 0/0 | 73/144 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Erythema (Any) (Skin and subcutaneous tissue disorders) | 65/123 | 44/144 | 0/0 | 0/0 | 0/0 | 0/0 | 43/134 — Infant Series Dose 3 / After Toddler Dose 3
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 80/152 | 19/151 | 0/0 | 63/139 | 51/106 | 39/137 | 0/0 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 83/142 | 50/150 | 0/0 | 65/144 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 57/123 | 40/143 | 0/0 | 0/0 | 0/0 | 0/0 | 36/133 — Infant Series Dose 3 / After Toddler Dose 3
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 22/148 | 3/152 | 0/0 | 14/136 | 24/102 | 10/134 | 0/0 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 43/134 | 10/147 | 0/0 | 19/140 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 24/120 | 8/139 | 0/0 | 0/0 | 0/0 | 0/0 | 13/131 — Infant Series Dose 3 / After Toddler Dose 3
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/148 | 0/151 | 0/0 | 0/135 | 0/98 | 0/133 | 0/0 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/133 | 0/147 | 0/0 | 0/138 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/118 | 0/138 | 0/0 | 0/0 | 0/0 | 0/0 | 0/130 — Infant Series Dose 3 / After Toddler Dose 3
Induration (Any) (Skin and subcutaneous tissue disorders) | 60/149 | 12/153 | 0/0 | 48/138 | 46/108 | 32/137 | 0/0 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose
Induration (Any) (Skin and subcutaneous tissue disorders) | 71/137 | 45/150 | 0/0 | 47/144 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Induration (Any) (Skin and subcutaneous tissue disorders) | 55/124 | 28/144 | 0/0 | 0/0 | 0/0 | 0/0 | 37/134 — Infant Series Dose 3 / After Toddler Dose 3
Induration (Mild) (Skin and subcutaneous tissue disorders) | 57/149 | 12/153 | 0/0 | 45/138 | 44/108 | 27/137 | 0/0 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose
Induration (Mild) (Skin and subcutaneous tissue disorders) | 68/137 | 43/150 | 0/0 | 43/143 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Induration (Mild) (Skin and subcutaneous tissue disorders) | 53/124 | 28/144 | 0/0 | 0/0 | 0/0 | 0/0 | 33/133 — Infant Series Dose 3 / After Toddler Dose 3
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 15/148 | 0/151 | 0/0 | 11/135 | 16/99 | 9/133 | 0/0 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 32/134 | 10/148 | 0/0 | 21/140 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 14/119 | 3/139 | 0/0 | 0/0 | 0/0 | 0/0 | 13/131 — Infant Series Dose 3 / After Toddler Dose 3
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/148 | 0/151 | 0/0 | 0/135 | 0/98 | 0/133 | 0/0 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/133 | 0/147 | 0/0 | 0/138 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/118 | 0/138 | 0/0 | 0/0 | 0/0 | 0/0 | 0/130 — Infant Series Dose 3 / After Toddler Dose 3
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 18/148 | 1/151 | 0/0 | 11/136 | 11/99 | 6/136 | 0/0 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 10/133 | 6/147 | 0/0 | 7/139 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 6/119 | 5/138 | 0/0 | 0/0 | 0/0 | 0/0 | 9/132 — Infant Series Dose 3 / After Toddler Dose 3
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 0/148 | 0/151 | 0/0 | 0/135 | 0/98 | 0/133 | 0/0 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 0/133 | 0/147 | 0/0 | 0/138 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 0/118 | 0/138 | 0/0 | 0/0 | 0/0 | 0/0 | 0/130 — Infant Series Dose 3 / After Toddler Dose 3
Fever ≥37.5°C but ≤39°C (General disorders) | 28/149 | 24/152 | 0/0 | 45/139 | 35/103 | 30/135 | 26/134 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose / After Toddler Dose
Fever ≥37.5°C but ≤39°C (General disorders) | 35/138 | 23/149 | 0/0 | 45/140 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Fever ≥37.5°C but ≤39°C (General disorders) | 23/120 | 21/141 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Fever>39°C but ≤40°C (General disorders) | 3/148 | 3/135 | 0/0 | 3/135 | 5/99 | 3/132 | 1/130 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose / After Toddler Dose
Fever>39°C but ≤40°C (General disorders) | 3/135 | 0/147 | 0/0 | 7/138 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Fever>39°C but ≤40°C (General disorders) | 2/118 | 1/138 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Fever >40.0°C (General disorders) | 0/148 | 0/151 | 0/0 | 0/135 | 1/98 | 0/132 | 0/130 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose / After Toddler Dose
Fever >40.0°C (General disorders) | 0/133 | 1/147 | 0/0 | 1/138 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Fever >40.0°C (General disorders) | 0/118 | 0/138 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Decreased appetite (General disorders) | 13/148 | 12/151 | 0/0 | 11/136 | 9/100 | 11/133 | 8/130 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose / After Toddler Dose
Decreased appetite (General disorders) | 16/135 | 8/147 | 0/0 | 15/138 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Decreased appetite (General disorders) | 10/119 | 9/138 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Irritability (General disorders) | 23/151 | 14/151 | 0/0 | 17/136 | 17/100 | 13/134 | 12/131 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose / After Toddler Dose
Irritability (General disorders) | 26/134 | 18/149 | 0/0 | 16/138 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Irritability (General disorders) | 12/118 | 10/139 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Increased sleep (General disorders) | 48/150 | 39/153 | 0/0 | 24/136 | 21/103 | 21/135 | 14/131 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose / After Toddler Dose
Increased sleep (General disorders) | 26/136 | 19/148 | 0/0 | 22/138 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Increased sleep (General disorders) | 19/119 | 26/141 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Decreased sleep (General disorders) | 25/151 | 23/151 | 0/0 | 16/136 | 11/101 | 10/133 | 9/131 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose / After Toddler Dose
Decreased sleep (General disorders) | 24/140 | 23/151 | 0/0 | 14/139 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Decreased sleep (General disorders) | 8/120 | 20/140 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Hives (urticaria) (General disorders) | 2/148 | 1/151 | 0/0 | 1/135 | 1/98 | 1/133 | 1/131 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose / After Toddler Dose
Hives (urticaria) (General disorders) | 4/133 | 0/147 | 0/0 | 3/138 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Hives (urticaria) (General disorders) | 2/119 | 0/138 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Use of antipyretic medication to treat symptoms (General disorders) | 2/148 | 2/151 | 0/0 | 8/136 | 4/98 | 6/133 | 2/130 — Infant Series Dose 1 / After Infant Series Dose 1 / Toddler Dose / After Toddler Dose
Use of antipyretic medication to treat symptoms (General disorders) | 3/134 | 3/147 | 0/0 | 7/138 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2 / After Infant Series Dose 2
Use of antipyretic medication to treat symptoms (General disorders) | 2/119 | 3/138 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.